CLINICAL TRIAL: NCT00098709
Title: A Randomized Clinical Trial of Fetal Pulse Oximetry
Brief Title: Fetal Pulse Oximetry Trial (FOX)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: The George Washington University Biostatistics Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HD36801-FOX; U10HD021410 (NIH); U10HD027869 (NIH); U10HD027917 (NIH); U10HD027860 (NIH); U10HD034116 (NIH); U10HD034208 (NIH); U10HD034136 (NIH); U10HD040500 (NIH); U10HD040485 (NIH); U10HD040544 (NIH); U10HD040545 (NIH); U10HD040560 (NIH); U10HD040512 (NIH); U10HD036801 (NIH)
Record Dates: First submitted 2004-12-07; First posted 2004-12-08 (Estimated); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Pregnancy
Keywords: pregnancy; labor, obstetric; fetal monitoring; oximetry; fetal heart rate; cardiotocography

INTERVENTIONS:
Device: Fetal pulse oximeter

SUMMARY:
The purpose of this study is to determine if the information provided to the physician by a fetal pulse oximeter during labor will reduce the chances of a cesarean delivery.

DETAILED DESCRIPTION:
Information on fetal well-being during labor is of great importance to the managing physician. The current use of the fetal heart rate monitor provides some information on fetal condition, and is the primary tool used to determine if immediate operative delivery is required. The fetal pulse oximeter can provide additional information regarding fetal oxygen saturation.

Intervention: A fetal oxygen saturation sensor is placed in the uterus, between the fetal cheek or forehead and the uterine wall. In half of the patients, the managing physician will have access to fetal oxygen saturation and fetal heart rate monitoring. In the other half of the patients, labor will be monitored by fetal heart rate alone.

Study hypothesis: The additional information provided by the use of the fetal pulse oximeter will reduce the chances of a cesarean delivery. The primary outcome is cesarean section for any indication and secondary outcomes are cesarean delivery for non-reassuring fetal heart rate or dystocia, and neonatal morbidity.

ELIGIBILITY:
Inclusion criteria:

* Nulliparous
* Singleton, cephalic pregnancy
* Gestational age at least 36 weeks, 0 days
* Cervical dilatation >= 2 cm
* Station -2 or below (5ths scale)
* Ruptured membranes
* Internal monitoring devices placed

Exclusion criteria:

* Need for immediate delivery
* Planned cesarean delivery
* Cervical dilatation > 6 cm
* Known fetal anomaly or demise
* Multifetal gestation
* Maternal fever
* Placenta previa
* Previous uterine surgery
* Active HSV infection
* Known HIV or hepatitis infection
* Diabetes requiring insulin
* Heart disease requiring medication
* Known chronic renal disease
* Enrollment in another labor study

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10000
Dates: Start 2002-05; Study Completion 2005-02

PRIMARY OUTCOMES:
cesarean delivery (any indication)

SECONDARY OUTCOMES:
cesarean delivery for non-reassuring fetal heart rate
cesarean delivery for dystocia
neonatal morbidity

CONTACTS AND LOCATIONS:
Overall Officials: Cathy Spong, MD, Study Director — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD); Elizabeth A Thom, Ph.D., Principal Investigator — George Washington University Biostatistics Center; Steven L Bloom, M.D., Study Chair — University of Texas
Locations (13):
- United States (13):
  - University of Alabama - Birmingham, Birmingham, Alabama
  - Northwestern University, Chicago, Illinois
  - Wayne State University, Detroit, Michigan
  - Columbia University, New York, New York
  - University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Case Western University, Cleveland, Ohio
  - Dexel University, Philadelphia, Pennsylvania
  - University of Pittsburgh Magee Womens Hospital, Pittsburgh, Pennsylvania
  - Brown University, Providence, Rhode Island
  - University of Texas - Southwest, Dallas, Texas
  - University of Texas - Houston, Houston, Texas
  - University of Utah Medical Center, Salt Lake City, Utah

REFERENCES:
- [Background] Goffinet F, Langer B, Carbonne B, Berkane N, Tardif D, Le Goueff F, Laville M, Maillard F. Multicenter study on the clinical value of fetal pulse oximetry. I. Methodologic evaluation. The French Study Group on Fetal Pulse Oximetry. Am J Obstet Gynecol. 1997 Nov;177(5):1238-46. doi: 10.1016/s0002-9378(97)70045-0. PMID 9396924
- [Background] Garite TJ, Dildy GA, McNamara H, Nageotte MP, Boehm FH, Dellinger EH, Knuppel RA, Porreco RP, Miller HS, Sunderji S, Varner MW, Swedlow DB. A multicenter controlled trial of fetal pulse oximetry in the intrapartum management of nonreassuring fetal heart rate patterns. Am J Obstet Gynecol. 2000 Nov;183(5):1049-58. doi: 10.1067/mob.2000.110632. PMID 11084540
- [Background] Bloom SL, Spong CY, Thom E, Varner MW, Rouse DJ, Weininger S, Ramin SM, Caritis SN, Peaceman A, Sorokin Y, Sciscione A, Carpenter M, Mercer B, Thorp J, Malone F, Harper M, Iams J, Anderson G; National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Fetal pulse oximetry and cesarean delivery. N Engl J Med. 2006 Nov 23;355(21):2195-202. doi: 10.1056/NEJMoa061170. PMID 17124017
- [Background] Rouse DJ, Weiner SJ, Bloom SL, Varner MW, Spong CY, Ramin SM, Caritis SN, Peaceman AM, Sorokin Y, Sciscione A, Carpenter MW, Mercer BM, Thorp JM Jr, Malone FD, Harper M, Iams JD, Anderson GD; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Second-stage labor duration in nulliparous women: relationship to maternal and perinatal outcomes. Am J Obstet Gynecol. 2009 Oct;201(4):357.e1-7. doi: 10.1016/j.ajog.2009.08.003. PMID 19788967
- [Background] Contag SA, Clifton RG, Bloom SL, Spong CY, Varner MW, Rouse DJ, Ramin SM, Caritis SN, Peaceman AM, Sorokin Y, Sciscione A, Carpenter MW, Mercer BM, Thorp JM Jr, Malone FD, Iams JD. Neonatal outcomes and operative vaginal delivery versus cesarean delivery. Am J Perinatol. 2010 Jun;27(6):493-9. doi: 10.1055/s-0030-1247605. Epub 2010 Jan 22. PMID 20099218
- [Background] Robinson BK, Mapp DC, Bloom SL, Rouse DJ, Spong CY, Varner MW, Ramin SM, Sorokin Y, Sciscione A, Mercer BM, Thorp JM Jr, Malone FD, Harper M, Ehrenberg H. Increasing maternal body mass index and characteristics of the second stage of labor. Obstet Gynecol. 2011 Dec;118(6):1309-1313. doi: 10.1097/AOG.0b013e318236fbd1. PMID 22105260
- [Background] Rouse DJ, Weiner SJ, Bloom SL, Varner MW, Spong CY, Ramin SM, Caritis SN, Grobman WA, Sorokin Y, Sciscione A, Carpenter MW, Mercer BM, Thorp JM Jr, Malone FD, Harper M, Iams JD, Anderson GD; Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) Maternal-Fetal Medicine Units Network (MFMU). Failed labor induction: toward an objective diagnosis. Obstet Gynecol. 2011 Feb;117(2 Pt 1):267-272. doi: 10.1097/AOG.0b013e318207887a. PMID 21252738
- [Background] Tita AT, Lai Y, Bloom SL, Spong CY, Varner MW, Ramin SM, Caritis SN, Grobman WA, Sorokin Y, Sciscione A, Carpenter MW, Mercer BM, Thorp JM Jr, Malone FD, Harper M, Iams JD. Timing of delivery and pregnancy outcomes among laboring nulliparous women. Am J Obstet Gynecol. 2012 Mar;206(3):239.e1-8. doi: 10.1016/j.ajog.2011.12.006. Epub 2011 Dec 16. PMID 22244471
- [Background] Segel SY, Carreno CA, Weiner SJ, Bloom SL, Spong CY, Varner MW, Rouse DJ, Caritis SN, Grobman WA, Sorokin Y, Sciscione A, Mercer BM, Thorp JM, Malone FD, Harper M, Iams JD; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Relationship between fetal station and successful vaginal delivery in nulliparous women. Am J Perinatol. 2012 Oct;29(9):723-30. doi: 10.1055/s-0032-1314895. Epub 2012 May 29. PMID 22644826
- [Background] Costantine MM, Lai Y, Bloom SL, Spong CY, Varner MW, Rouse DJ, Ramin SM, Caritis SN, Peaceman AM, Sorokin Y, Sciscione A, Mercer BM, Thorp JM, Malone FD, Harper M, Iams JD; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Population versus customized fetal growth norms and adverse outcomes in an intrapartum cohort. Am J Perinatol. 2013 Apr;30(4):335-41. doi: 10.1055/s-0032-1324708. Epub 2012 Aug 14. PMID 22893556
- [Background] Langen ES, Weiner SJ, Bloom SL, Rouse DJ, Varner MW, Reddy UM, Ramin SM, Caritis SN, Peaceman AM, Sorokin Y, Sciscione A, Carpenter MW, Mercer BM, Thorp JM Jr, Malone FD, Iams JD; Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) Maternal-Fetal Medicine Units (MFMU) Network. Association of Cervical Effacement With the Rate of Cervical Change in Labor Among Nulliparous Women. Obstet Gynecol. 2016 Mar;127(3):489-495. doi: 10.1097/AOG.0000000000001299. PMID 26855099
- See also: The public website of the NICHD Maternal Fetal Medicine Units (MFMU) Network — http://www.bsc.gwu.edu/mfmu/